CLINICAL TRIAL: NCT06035952
Title: Prospective Validation of 3D Body Surface Modeling for Patient Monitoring in Adolescent Idiopathic Scoliosis
Brief Title: Study of 3D Scanning for Adolescent Scoliosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NSite Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 54101
Record Dates: First submitted 2023-08-31; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Scoliosis
Keywords: scoliosis; topographical scanning
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Intervention: This study will have one cohort. This group of patients will undergo 3D scanning with a smartphone, and will also have standard of care diagnostics, such as an X-ray.
  Interventions: Diagnostic Test: 3D topographical scan

INTERVENTIONS:
Diagnostic Test: 3D topographical scan — Subjects will undergo a quick, radiation-free, no contact 3D scan using a smartphone.

SUMMARY:
The investigators aim to validate three-dimensional topographical scanning technology as a tool for evaluation of scoliosis. Through the incorporation of 3D topographical technology in the measurement of deformity, the investigators hope to validate a novel approach to quantify deformity progression and provide an accessible alternative to traditional radiographic workup.

DETAILED DESCRIPTION:
The study design will be prospective observational. Patients 10 to 18 years old being evaluated or followed for scoliosis will be included. Those unable to complete the consent and assent processes will not be enrolled. Members of the research team will review the clinic schedule through EPIC each week to identify eligible patients. Member of the patient's care team, such as the physician, will introduce the study to the patient. If the patient and the patient's caregivers are interested in learning more and/or participating, a member of the research team will provide study-related information and obtain informed consent via written or electronic consent, assent, and, if necessary, short form consent.

If a patient consents to participate, members of the research team will conduct the 3D topographical scan in a private room in the clinic. This involves 360 degree scans using a smartphone camera. Participants will also receive any standard of care x-rays during the visit. The investigators will then analyze the ability of the 3D smartphone scan to estimate the Cobb Angle measured on the X-ray, to infer the magnitude of the scoliosis deformity.

ELIGIBILITY:
Inclusion Criteria:

* Ages 10 and 18 years old

Exclusion Criteria:

* Scoliosis caused by another condition (e.g., secondary scoliosis)
* Parents/guardians unable to consent
* English is not the primary language (to avoid miscommunication)

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population will include children and adolescent patients 10 to 18 years old who present to a pediatric orthopedic clinic for scoliosis evaluation. This age range was chosen as it is the age range in which Adolescent Idiopathic Scoliosis commonly appears, and the device is intended for screening for this condition.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Accuracy of scanning device to predict clinically significant Cobb Angle | Through study completion, an average of 3 months
  The primary study endpoint, or primary outcome, is whether the 3D scan's predicted probability of clinically significant Cobb angle correlates with the ground truth radiograph obtained Cobb angle at the defined rate. The percentage (%) of patient scans with predicted probabilities that correlate with ground truth results will be reported.

SECONDARY OUTCOMES:
Repeatability of 3D scan analysis | Within 48 hours
  After the 3D scan is obtained, several personnel will align the scan relative to grid coordinates, and place a region of interest on the back of the scan. Measurements will be performed which will generate an asymmetry value, which is used to assess Cobb Angle correlation. The investigators will determine the repeatability of this manual scan assessment process.

CONTACTS AND LOCATIONS:
Overall Officials: Kali Tileston, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Palo Alto, California
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No